CLINICAL TRIAL: NCT00875641
Title: Safety Study of GSK Biologicals' Rotarix® (Rotavirus Vaccine, Live, Oral) Administered to a Birth Cohort in United States Health Insurance Plans
Brief Title: Safety Study of GSK Biologicals' Rotavirus Vaccine (Rotarix®) Administered to Children Aged <1 Year in the United States
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112229
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-06

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HRV cohort: HRV (Human Rotavirus) cohort consisted of infants aged less than 1 year, enrolled in the participating health insurance plans within 30 days of birth and who received at least one dose of Rotarix vaccination as part of their normal health care (with no previous dose of RotaTeq prior to or concurrent with the first Rotarix vaccination).
  Interventions: Other: Health Insurance Database
- Concurrent Control cohort: Concurrent control cohort consisted of infants aged less than 1 year, enrolled in the participating health insurance plans, who were contemporaneous with the Rotarix vaccinees and who received at least one dose of IPV (Inactivated Poliovirus vaccine) with or without RotaTeq vaccination (with no previous dose of Rotarix prior to or concurrent with the first IPV vaccination).
  Interventions: Other: Health Insurance Database
- Recent Historical Control cohort: Recent historical control cohort consisted of infants aged less than 1 year of age, enrolled in participating health insurance plans, vaccinated with at least one dose of IPV (Inactivated Poliovirus vaccine) between 1 January 2004 (OptumInsight) or 1 January 2006 (HealthCore) and 31 July 2008 and who did not receive any dose of rotavirus vaccination during the study period.
  Interventions: Other: Health Insurance Database

INTERVENTIONS:
Other: Health Insurance Database — Review of two health insurance databases in the US to determine the safety outcomes among infants who have received Rotarix or IPV vaccination.

SUMMARY:
This observational cohort study, conducted through two existing large administrative health databases in the US (outside the Vaccine Safety Datalink) is planned to confirm the safety profile regarding lack of any association of intussusception with Rotarix within 60 days of vaccination in a real life setting (routine use) in the US. This study will also include monitoring of Kawasaki disease, convulsions, hospitalizations due to acute lower respiratory tract infections and all-cause deaths within 60-days of vaccination.

This study involves three cohorts, one exposed and two control cohorts: infants who receive Rotarix (Exposed cohort) and infants who receive IPV vaccination (Unexposed cohort A and B).

This is a combined prospective and retrospective cohort study. Prospective component of the study identifies and compares study outcomes following Rotarix and IPV vaccination in the Exposed cohort and Unexposed cohort A, respectively.

Retrospective component of the study identifies and compares study outcomes following IPV vaccination in the Unexposed cohort B.

ELIGIBILITY:
Inclusion Criteria:

For Exposed cohort:

* Infants aged less than 1 year at study entry.
* Infants who are enrolled in one of the two participating health insurance plans databases within 30 days of birth.
* Have complete medical coverage and pharmacy benefits.
* Received at least one dose of Rotarix from 1 August 2008.
* Infants receiving Rotarix liquid formulation will also be eligible.

For Unexposed cohort A:

* Infants aged less than 1 year at study entry.
* Infants who are enrolled in one of the two participating health insurance plans databases within 30 days of birth.
* Have complete medical coverage and pharmacy benefits.
* Received at least one dose of IPV vaccine from 1 August 2008, with or without RotaTeq vaccination.
* Frequency-matched to the Rotarix cohort by gender, age at first vaccination (±1 week) and calendar quarter of vaccination within the same year.

For Unexposed cohort B:

* Infants who are enrolled in one of the two participating health insurance plans databases within 30 days of birth.
* Had complete medical coverage and pharmacy benefits.
* Received at least one dose of IPV vaccine.
* Vaccinated between 1 January 2006 (inclusive) and 31 July 2008 (inclusive).
* Not received any dose of rotavirus vaccination.
* Frequency-matched to the Rotarix cohort by gender, age at first vaccination (±1 week) and calendar quarter of vaccination.

Exclusion Criteria:

For Exposed cohort:

• Subject has received any dose of RotaTeq prior to the first Rotarix vaccine during the study period.

For Unexposed cohort A:

• Subject has received any dose of Rotarix prior to the first IPV vaccine during the study period.

For Unexposed cohort B:

• Subject has received any dose of rotavirus vaccines prior to the first IPV vaccine.

Max Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children affiliated to two participating health insurance plans.
Sampling Method: Non-Probability Sample
Enrollment: 390659 (Actual)
Dates: Start 2009-04-20 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were identified through the automated corresponding health insurance plan databases, OptumInsight Life Sciences Research Database (from United Healthcare) and the HealthCore Integrated Research Database (HIRDSM) (part of Anthem, formerly known as WellPoint).
Period: Overall Study
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Started | 57931 | 173384 | 159344
Completed | 57931 | 173384 | 159344
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort | Total
Number analyzed (Participants) | 57931 | 173384 | 159344 | 390659
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.0 (0.7) | 2.0 (0.7) | 2.0 (0.7) | 2.0 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27929 | 83528 | 77128 | 188585
  Male | 30002 | 89856 | 82216 | 202074
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  US Geographic Region: Northeast | 8461 | 18093 | 22171 | 48725
  US Geographic Region: South/Southeast | 19875 | 59167 | 61965 | 141007
  US Geographic Region: Midwest | 17101 | 51046 | 41114 | 109261
  US Geographic Region: West | 12494 | 45078 | 34094 | 91666

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rates of Intussusceptions (IS) Among the HRV Cohort and Comparator Cohorts
Description: Incidence rates were calculated following the first 2 doses of study vaccine as the number of events divided by the sum of the person-time in that risk period. Person-time was defined as the number of days at risk for the study outcomes. Person-time was calculated in months by dividing the number of person-days by (365.25/12).
Time Frame: 60 days following each vaccination
Population: Analysis was performed on study population comprising of birth cohorts affiliated with 2 participating health insurance plans, United Healthcare & WellPoint, which were eligible for rotavirus vaccination according to routine recommendations. Within this population of infants, HRV, Concurrent Control & Recent Historical Control cohorts were defined.
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-59 days, Any Dose | 0.021 [0.006 to 0.055] | 0.022 [0.012 to 0.037] | 0.021 [0.010 to 0.037]
  0-59 days, Dose 1 | 0.028 [0.006 to 0.082] | 0.012 [0.003 to 0.032] | 0.017 [0.006 to 0.040]
  0-59 days, Dose 2 | 0.013 [0.000 to 0.070] | 0.032 [0.015 to 0.061] | 0.025 [0.009 to 0.054]

2. Primary Outcome: Incidence Rates of IS Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 7 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-6 days, Any Dose | 0.000 [0.000 to 0.161] | 0.014 [0.000 to 0.075] | 0.000 [0.000 to 0.056]
  0-6 days, Dose 1 | 0.000 [0.000 to 0.278] | 0.000 [0.000 to 0.093] | 0.000 [0.000 to 0.101]
  0-6 days, Dose 2 | 0.000 [0.000 to 0.383] | 0.029 [0.001 to 0.162] | 0.000 [0.000 to 0.124]

3. Primary Outcome: Incidence Rates of IS Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 30 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-29 days, Any Dose | 0.010 [0.000 to 0.058] | 0.026 [0.011 to 0.050] | 0.022 [0.008 to 0.047]
  0-29 days, Dose 1 | 0.000 [0.000 to 0.066] | 0.006 [0.000 to 0.033] | 0.020 [0.004 to 0.057]
  0-29 days, Dose 2 | 0.025 [0.001 to 0.137] | 0.048 [0.019 to 0.099] | 0.024 [0.005 to 0.070]

4. Secondary Outcome: Incidence Rates of Kawasaki Disease Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 60 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-59 days, Any Dose | 0.000 [0.000 to 0.020] | 0.008 [0.003 to 0.019] | 0.009 [0.003 to 0.022]
  0-59 days, Dose 1 | 0.000 [0.000 to 0.034] | 0.006 [0.001 to 0.023] | 0.014 [0.004 to 0.035]
  0-59 days, Dose 2 | 0.000 [0.000 to 0.046] | 0.011 [0.002 to 0.031] | 0.004 [0.000 to 0.023]

5. Secondary Outcome: Incidence Rates of Convulsions Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 60 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-59 days, Any Dose | 0.230 [0.166 to 0.310] | 0.142 [0.113 to 0.175] | 0.146 [0.116 to 0.183]
  0-59 days, Dose 1 | 0.252 [0.166 to 0.366] | 0.121 [0.086 to 0.166] | 0.124 [0.087 to 0.171]
  0-59 days, Dose 2 | 0.200 [0.115 to 0.326] | 0.165 [0.121 to 0.220] | 0.174 [0.125 to 0.235]

6. Secondary Outcome: Incidence Rates of Acute Lower Respiratory Tract Infection (LRTI) Hospitalisation Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 60 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-59 days, Any Dose | 1.518 [1.346 to 1.705] | 1.320 [1.230 to 1.415] | 1.669 [1.561 to 1.782]
  0-59 days, Dose 1 | 1.696 [1.459 to 1.962] | 1.529 [1.397 to 1.671] | 2.008 [1.848 to 2.177]
  0-59 days, Dose 2 | 1.278 [1.042 to 1.551] | 1.079 [0.961 to 1.208] | 1.260 [1.123 to 1.410]

7. Secondary Outcome: Incidence Rates of Acute LTRI Hospitalisation Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 7 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-6 days, Any Dose | 1.397 [0.955 to 1.972] | 0.932 [0.725 to 1.180] | 1.406 [1.135 to 1.722]
  0-6 days, Dose 1 | 1.960 [1.280 to 2.871] | 1.184 [0.870 to 1.575] | 1.921 [1.497 to 2.427]
  0-6 days, Dose 2 | 0.622 [0.228 to 1.354] | 0.641 [0.401 to 0.970] | 0.774 [0.491 to 1.162]

8. Secondary Outcome: Incidence Rates of Acute LTRI Hospitalisation Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 30 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-29 days, Any Dose | 1.593 [1.351 to 1.865] | 1.383 [1.255 to 1.519] | 1.788 [1.634 to 1.952]
  0-29 days, Dose 1 | 1.858 [1.518 to 2.252] | 1.523 [1.341 to 1.721] | 2.166 [1.939 to 2.412]
  0-29 days, Dose 2 | 1.228 [0.911 to 1.619] | 1.221 [1.048 to 1.414] | 1.327 [1.132 to 1.544]

9. Secondary Outcome: Incidence Rates of All-cause Mortality Among the HRV Cohort and Comparator Cohorts
Description: as for outcome 1
Time Frame: 60 days following each vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidences/Person-Month
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
Number analyzed (Participants) | 57931 | 173384 | 159344
Incidences/Person-Month
  0-59 days, Any Dose | 0.048 [0.022 to 0.091] | 0.045 [0.030 to 0.065] | 0.062 [0.043 to 0.087]
  0-59 days, Dose 1 | 0.047 [0.015 to 0.109] | 0.059 [0.036 to 0.092] | 0.075 [0.047 to 0.114]
  0-59 days, Dose 2 | 0.050 [0.014 to 0.128] | 0.029 [0.012 to 0.057] | 0.045 [0.023 to 0.081]

ADVERSE EVENTS:
Arm/Group | HRV Cohort | Concurrent Control Cohort | Recent Historical Control Cohort
All-Cause Mortality (participants affected / at risk) | 9/57931 | 27/173384 | 33/159344
Serious Adverse Events (participants affected / at risk) | 0/57931 | 0/173384 | 0/159344
Other Adverse Events (participants affected / at risk) | 0/57931 | 0/173384 | 0/159344

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.